CLINICAL TRIAL: NCT07273695
Title: Assessing Real Life Effectiveness of Treatment in Neurodevelopmental Disorders
Acronym: ALERT
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 1120; Ricerca Corrente (Other Grant/Funding Number: Italian Ministry og Health)
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Emotional Dysregulation; Externalizing Problems; Oppositional Defiant; Conduct Disorder; Disruptive Behaviours; Attention Deficit Hyerpactivity Disorder
Keywords: attention deficit hyperactivity disorder; child training; methylphenidate; emotional dysregulation; externalizing disorders/behaviors
MeSH Terms: conditions — Conduct Disorder; Attention Deficit Disorder with Hyperactivity; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- participants beguinning drug treatment: children and adolescents with emotional dysregulation, externalizing disorders and/or ADHD beguinning drug treatment (MPH)
  Interventions: Drug: methyphenidate
- participants beguinning group psychotherapy: children and adolescents with emotional dysregulation externalizing disorders and/or ADHD beguinning group psychotherapy (child training)
  Interventions: Behavioral: Group psychological treatment
- control groups: children and adolescents with emotional dysregulation, externalizing disorders and/or ADHD in waiting list to beguin their treatment

INTERVENTIONS:
Drug: methyphenidate — According to clinical practice and national guidelines, subjects who meet the severity criteria and who express their consent to undertake pharmacological therapy undergo the medical tests required for the initiation of therapy. Only subsequently, according to standard clinical practice, the patient is subjected to the test dose of methylphenidate in the facility, in order to monitor any side effects. The dosage prescribed to patients varies depending on the subject's characteristics (5-20 mg/day) and is set by the child neuropsychiatrist based on the response to treatment, tolerability, and adverse effects, , according to Italian clinical guidelines for children and adolescents (SINPIA, 2002).
  Other Names: Drug treatment
  Groups: participants beguinning drug treatment
Behavioral: Group psychological treatment — The treatment consists of 16 weekly sessions lasting 1.5 hours. The total duration of the intervention is 4 months for a total of 16 sessions. The therapeutic group will be a closed group with approximately 6 patients per group. Patients will be assigned to different groups based on age and skills (8-11 and 12-15 years).
  The proposed interventions are based on the theoretical principles and techniques of Schema Therapy for developmental age (Christof Loose, Peter Graaf, Gerhard Zarbock & Ruth A. Holt; Italian edition edited by Stefano Terenzi and Rosario Capo, 2013) or Acceptance and Commitment Therapy (Vanzin et al., 2020a; 2020b) for externalizing disorders.
  Groups: participants beguinning group psychotherapy

SUMMARY:
The goal of this observational study is to learn if and how pharmacological and psychotherapeutic group treatments can treat clinical symptoms of children and adolescent patients with ADHD.

The main questions it aims to answer are:

* Are pharmacological and psychotherapeutic treatments effective on the clinical symptoms of patients with ADHD?
* Are pharmacological and psychotherapeutic treatments effective on symptoms of emotion-behavioral dysregulation?
* Is it possible to find associations between individual characteristics and treatment responses evaluating behavioral and neural correlates in children and adolescents with traits of emotion-behavioral dysregulation, externalizing disorders, and/or ADHD, using a panel of multimodal measures. May the data collected contribute to the definition of profiles useful for generating predictive hypotheses aimed at developing more personalized interventions?

Researchers will compare the data collected from patients treated with pharmacological and psychotherapeutic group treatments with the data of subjects of comparable sex/gender, age, diagnoses, on the waiting list for treatment to see if pharmacological and psychotherapeutic treatments effects ADHD and emotional dysregulation symprtoms.

Participants, patients who are offered treatment by clinicians according to standard clinical practice, will be asked to participate in the study by undergoing experimental assessments before and after the treatment.

The multimodal panel of proposed assessments includes:

* behavioral assessments, conducted through the completion of clinical and socio-demographic questionnaires;
* neuropsychological assessments, conducted through standardized computerized neuropsychological tests;
* neurophysiological assessments, conducted through the recording of NIRS (near infrared spectroscopy) and EEG (electroencephalogram) signals during an attentional task (Go-NoGo) and via a smartwatch.

DETAILED DESCRIPTION:
Study Objectives The research protocol involves a multimodal assessment of participants before and after various types of treatment. The ultimate goal is to evaluate the effectiveness of treatment on symptoms of emotion-behavioral dysregulation, externalizing disorders, and/or ADHD. This is done by analyzing the multimodal data collected before treatment. This allows us to predict treatment effectiveness and propose a more personalized and targeted intervention for each patient.

Primary Objective To evaluate the effectiveness of pharmacological and psychotherapeutic treatments on the clinical symptoms of patients with ADHD.

Secondary Objective To evaluate the effectiveness of pharmacological and psychotherapeutic treatments for symptoms of emotion-behavioral dysregulation.

Exploratory Objective To evaluate behavioral and neural correlates in preadolescents and adolescents with traits of emotional-behavioral dysregulation, externalizing disorders, and/or ADHD, using a panel of multimodal measures, in order to explore possible associations between individual characteristics and treatment responses. The data collected may contribute to the definition of profiles useful for generating predictive hypotheses, to be validated in subsequent studies, aimed at developing more personalized interventions.

Study Design The objectives will be pursued within a multicenter, non-profit, prospective and retrospective interventional study, non-randomized and non-blinded.

Patients who are offered treatment by clinicians, according to standard clinical practice, will be asked to participate in the study by undergoing experimental assessments before and after treatment.

Specifically, patients with symptoms of emotional-behavioral dysregulation, externalizing disorders, and/or ADHD will be recruited and offered multiple assessment sessions over a 9-12-month period (depending on the treatment assigned according to clinical practice).

Controls will also be recruited: subjects of comparable gender and age, diagnosed with externalizing disorders, ADHD, and/or symptoms of emotional dysregulation who are on the treatment waiting list. They will be offered the same assessments but will not receive any treatment.

Recruitment began in September 2025 and continue until October/November 2026. The study will conclude in December 2026.

The treatments that will be offered to the patients evaluated within this project are of a variety of nature: 1)group psychoeducation and psychotherapy interventions aimed at preadolescents and adolescents; 2) treatments with psychotropic drugs.

Pre-treatment assessments will include:

Socio-demographic and clinical behavioral characterization with questionnaires administered to parents/caregivers of participants and to the participants themselves (based on the participants' age); Clinical neuropsychological characterization with computerized tasks to assess attention, inhibition, and flexibility; Characterization of hemodynamic and electrical activity during attention tasks using near-infrared spectroscopy (NIRS) and electroencephalogram (EEG); Characterization of the physiological profile through the acquisition of data deriving from sympathetic nervous system activation and movement, using a Samsung Galaxy Watch5 smartwatch.

Three follow-ups will be offered:

Subsample receiving group psychological intervention or on a waiting list:

T1: at the first treatment session; T2: at the end of treatment (after 16 weeks); T3: 6 months after the end of treatment.

Pharmacotherapy subsample:

T1: at the same time as the drug test dose; T2: at the end of the drug titration phase (after 8-12 weeks of continuous treatment); T3: 6 months after the end of titration.

Study Population Sixty patients with symptoms of emotional behavioral dysregulation, externalizing disorders, and ADHD will be recruited at referral centers in Lombardy (the UONPIA of the ASST Brianza and the IRCCS Eugenio Medea - Bosisio Parini site) and Veneto (the IRCCS Eugenio Medea - Conegliano site). Each center is expected to recruit 20 patients for treatment.

Twenty controls (waiting list patients) will also be recruited: subjects of comparable age, sex, and gender, with comparable symptomatology who are not undergoing any treatment.

Behavioral assessments will be conducted through the completion of clinical and socio-demographic questionnaires at each recruitment center.

Neuropsychological (ANT) and neurophysiological (NIRS, EEG, smartwatch) assessments will be conducted at the IRCCS MEDEA.

Treatments will be administered at each recruiting center: pharmacological treatments will be administered at the IRCCS E Medea facilities, while psychological treatments will be administered at all participating centers.

The data will be analyzed by researchers at IRCCS Eugenio Medea, ASST Brianza, and the Iluria company. Iluria Ltd. is a digital health company specializing in ADHD. Iluria Ltd. will analyze neurophysiological data collected with the Samsung Galaxy Watch5 smartwatch. For details, see the section "Study Endpoints - Neurophysiological Measures."

Eligibility Criteria Patients with symptoms of emotional-behavioral dysregulation, externalizing disorders, and/or ADHD will be recruited. According to clinical practice, the presence of these symptoms and diagnoses must be assessed prior to enrollment in the research project by experienced clinicians (psychologists, psychotherapists, and child neuropsychiatrists) through clinical interviews and diagnostic tools (questionnaires, interviews).

Children and adolescents aged 8-15 will be recruited. For psychotherapeutic treatment, participants will be divided into separate groups based on age and skills: 8-11 and 12-15 years old.

Patients with an IQ greater than 75 will be recruited, and, for the psychotherapeutic treatment group, those with good mentalization skills.

Pharmacological intervention will be offered in cases indicated, following international guidelines (for example, for ADHD, treatment with methylphenidate is administered in cases of Clinical Global Index severity (CGI-S) ≥ 4).

A control group will be recruited, consisting of patients on the treatment waiting list with the same diagnoses and comparable age. They will be administered the same clinical, neuropsychological, behavioral, and neurophysiological protocol. No post-clinical treatment will be offered, and no waiting list will be extended to complete the assessments included in the research protocol.

Interventions Intervention A

Treatments proposed based on clinical practice and national guidelines:

1. Psychological Group Treatment The treatment consists of 16 weekly sessions lasting 1.5 hours. The total duration of the intervention is 4 months for a total of 16 sessions. The therapeutic group will be a closed group with approximately 6 patients per group. Patients will be assigned to different groups based on age and skills (8-11 and 12-15 years).

   The proposed interventions are based on the theoretical principles and techniques of Schema Therapy for Developmental Age or Acceptance and Commitment Therapy for externalizing disorders.
2. Pharmacological Treatment Following clinical observation by the child neuropsychiatrist and upon reaching the severity threshold (≥ 4) on the CGI-S scale, meeting the criteria for pharmacological treatment according to national guidelines (SINPIA, 2002), the subjects will be prescribed methylphenidate, an active ingredient commonly used in first-line medications for ADHD. According to clinical practice and national guidelines, subjects who meet the severity criteria and who consent to pharmacological therapy undergo the required medical examinations for initiation of therapy. Only subsequently, according to standard clinical practice, is the patient administered a test dose of methylphenidate in the facility to monitor for any side effects. The dosage prescribed to patients varies depending on the individual's characteristics (5-20 mg/day) and is set by the child neuropsychiatrist based on treatment response, tolerability, and adverse effects, in accordance with Italian clinical guidelines for children and adolescents (SINPIA, 2002).

Intervention B (e.g., comparison) The same assessments (reported in the "Data Collection" section at T0, T2, and T3, with the same time intervals reported in the "Study Timeline" section) are also administered to the control group, which is not subjected to any type of treatment, in order to evaluate the learning effect of the neuropsychological tasks and the temporal variation in psychopathological traits not due to the intervention.

Clinical measures: Conners Rating Scales 3 questionnaires; Child Behavior CheckList for ages 6-18 - CBCL/6-18; Youth Self-Report for ages 11-18 - YSR/11-18; Difficulties in Emotion Regulation Scale - DERS; Parent Problem Checklist; Relationship Quality Index; The proposed Dyadic Adjustment Scale; Clinical Global Assessment Scale, C-GAS; Clinical Global Impressions Severity Scale, CGI-S; Clinical Global Impressions Improvement Scale, CGI-S. neuropsychological assessments (Amsterdam Neuropsychological Task - ANT) are standardized instruments for age and gender. The resulting measures will be aggregated as group means and compared both with the standardized means expected for that sample, in order to characterize the sample before the start of treatment, and as repeated measures for each sample to assess the change over time resulting from the proposed intervention. The evaluation of the change resulting from the interventions will be assessed at both T2 and T3.

Neurophysiological measures: measures derived from NIRS, EEG, and smartwatch acquisitions will be preprocessed to eliminate Artifacts. Preprocessing measures will be aggregated as group averages and compared across groups to characterize the sample before treatment begins. In this analysis, data previously collected in a group of typically developing children and adolescents provide a baseline for fNIRS and EEG assessments. Furthermore, these data will be analyzed as repeated measures for each sample to assess the change over time resulting from the proposed intervention. Change resulting from the interventions will be assessed at both T2 and T3. Measures acquired at T0 and T1 will be used to predict T2 and T3 measures.

Socio-demographic and risk factor measures: these measures will be included as covariates or predictors in models predicting change in clinical and neurophysiological measures resulting from treatments.

Study Design Study Timeline T0 - Once diagnostic assessments are completed according to clinical practice, participants will be assessed before treatment begins; T1 - Participants treated with Participants receiving pharmacotherapy will be assessed on the day they first start taking the medication; participants receiving group psychotherapy will be assessed at their first meeting; T2 - Participants receiving pharmacotherapy will be assessed three months after starting treatment or at the end of the drug titration phase; participants receiving group psychotherapy will be assessed at the end of the intervention; T3 - 6 months after T2.

ELIGIBILITY:
Inclusion Criteria

* Children and adolescents aged 8-15 years;
* Diagnosis of externalizing disorder, ADHD, and/or emotional dysregulation (assessed with questionnaires, interviews, and/or clinical observation);
* Intelligence quotient ≥ 75.

Exclusion Criteria

* IQ < 75;
* Substance abuse and addictions;
* Psychosis;
* Acute disorders;
* Organic brain disorders;
* Presence of neurological diseases, epilepsy;
* Genetic syndromes;
* Co-diagnosis with other psychiatric or neurodevelopmental disorders (e.g., autism, anxiety, depression, etc.) and prior psychopharmacological therapy will not be considered exclusion criteria but will be recorded and declared.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with symptoms of emotional-behavioral dysregulation, externalizing disorders, and/or ADHD will be recruited. The presence of these symptoms and diagnoses must be assessed prior to entry into the research project by experienced clinicians through clinical interviews and questionnaires.
  Children and adolescents aged 8-15 will be recruited. For psychotherapeutic treatment, participants will be divided into separate groups based on age and skills: 8-11 and 12-15.
  Patients with an IQ greater than 75 will be recruited, and, for the psychotherapeutic treatment group, those with good mentalization skills.
  Pharmacological intervention will be proposed in indicated cases following international guidelines (for example, for ADHD, treatment with methylphenidate is administered in cases of Clinical Global Index severity (CGI-S) ≥ 4).
  A control group will be recruited consisting of patients on the waiting list for treatment, with the same diagnoses and comparable age.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impressions - Severity Scale | T2 (2-3 months), T3 (6 months)
  Clinical improvement measured with CGI-s (Clinical Global Impression - severity)(minimum value: 1 = "normal, not ill"; maximun value: 7 = "very severely ill" )

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale - DERS | T2 (2-3 months), T3 (6 months)
  Questionnaire, total score, t scores

OTHER OUTCOMES:
explanatory outcomes | T2 (2-3 months), T3 (6 months)
  functional Near Infrared Spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Maria Nobile, PhD, MD, Principal Investigator — IRCCS E Medea Scientific Institute
Locations (1):
- IRCCS E Medea Scientific Institute - Asssociazione La Nostra Famiglia, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: Undecided
pseudonymized data will be shared under request via zenodo

REFERENCES:
- [Background] Mauri M, Grazioli S, Crippa A, Bacchetta A, Pozzoli U, Bertella S, Gatti E, Maggioni E, Rosi E, Diwadkar V, Brambilla P, Molteni M, Nobile M. Hemodynamic and behavioral peculiarities in response to emotional stimuli in children with attention deficit hyperactivity disorder: An fNIRS study. J Affect Disord. 2020 Dec 1;277:671-680. doi: 10.1016/j.jad.2020.08.064. Epub 2020 Sep 1. PMID 32911217
- [Background] Achenbach, T. (2001). Manual for the ASEBA school-age forms and profiles
- [Background] Vanzin, L., Mauri, V., Valli, A., Pozzi, M., Presti, G., Oppo, A., ... & Nobile, M. (2020a). Clinical effects of an ACT-group training in children and adolescents with attention-deficit/hyperactivity disorder. Journal of Child and Family Studies, 29, 1070-1080.
- [Background] Vanzin, L., Crippa, A., Mauri, V., Valli, A., Mauri, M., Molteni, M., & Nobile, M. (2020b). Does ACT-group training improve cognitive domain in children with attention deficit hyperactivity disorder? A single-arm, open-label study. Behaviour Change, 37(1), 33-44. doi:https://doi.org/10.1017/bec.2020.3
- [Background] Conners C. K. (2008), Conners 3rd Edition (Conners 3). Ad. it. di C. Primi e D. Maschietto, Giunti Psychometrics, Firenze 2017.
- [Background] Mauri M, Crippa A, Bacchetta A, Grazioli S, Rosi E, Gazzola E, Gallace A, Nobile M. The utility of NIRS technology for exploring emotional processing in children. J Affect Disord. 2020 Sep 1;274:819-824. doi: 10.1016/j.jad.2020.06.004. Epub 2020 Jun 3. PMID 32664020
- [Background] Grazioli S, Mauri M, Crippa A, Maggioni E, Molteni M, Brambilla P, Nobile M. Light up ADHD: II. Neuropharmacological effects measured by near infrared spectroscopy: is there a biomarker? J Affect Disord. 2019 Feb 1;244:100-106. doi: 10.1016/j.jad.2018.10.100. Epub 2018 Oct 9. PMID 30332620
- [Background] Grazioli S, Rosi E, Mauri M, Crippa A, Tizzoni F, Tarabelloni A, Villa FM, Chiapasco F, Reimers M, Gatti E, Bertella S, Molteni M, Nobile M. Patterns of Response to Methylphenidate Administration in Children with ADHD: A Personalized Medicine Approach through Clustering Analysis. Children (Basel). 2021 Nov 4;8(11):1008. doi: 10.3390/children8111008. PMID 34828721
- [Background] Mauri M, Nobile M, Bellina M, Crippa A, Brambilla P. Light up ADHD: I. Cortical hemodynamic responses measured by functional Near Infrared Spectroscopy (fNIRS): Special Section on "Translational and Neuroscience Studies in Affective Disorders" Section Editor, Maria Nobile MD, PhD. This Section of JAD focuses on the relevance of translational and neuroscience studies in providing a better understanding of the neural basis of affective disorders. The main aim is to briefly summarise relevant research findings in clinical neuroscience with particular regards to specific innovative topics in mood and anxiety disorders. J Affect Disord. 2018 Jul;234:358-364. doi: 10.1016/j.jad.2017.11.087. Epub 2017 Nov 21. PMID 29195758